CLINICAL TRIAL: NCT01372904
Title: Prevention of Cisplatin-Induced Hearing Loss by Intratympanic Dexamethasone Treatment.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CIS 4/2011
Record Dates: First submitted 2011-06-13; First posted 2011-06-14 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Cisplatin Ototoxicity
Keywords: Cisplatin; Hearing loss; Ototoxicity; Intratympanic injection; Dexamethasone; Steroids; Prevention
MeSH Terms: conditions — Hearing Loss; Ototoxicity | interventions — dexamethasone 21-phosphate; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dexamethasone (Experimental)
  Interventions: Drug: Dexamethasone Phosphate

INTERVENTIONS:
Drug: Dexamethasone Phosphate — 0.7ml of Dexamethasone Phosphate 10mg/ml would be injected unilaterally to the middle ear using 25 gauge spinal needle.
  The trans-tympanic membrane injection would take place at the posterior inferior quadrant of the ear drum facing the round window niche. The patient would be instructed to lie down for 20 minutes after the injection with the treated side up and to avoid swallowing or coughing. Intratympanic Dexamethasone would be delivered immediately prior to each cisplatin treatment as maximal level.
  Other Names: Decadron, Dexamethasone Intensol, Dexpak Taperpak, Zema Pak

SUMMARY:
Cisplatin is a widely used chemotherapeutic agent for the treatment of various malignant neoplasms, including testicular, ovarian, bladder, cervix uteri, head and neck and lung cancers.

One of the common side-effects of this drug is bilateral, symmetric, progressive and usually irreversible sensorineural hearing loss.

Cisplatin induces cochlear toxicity by the production of reactive oxygen species (ROS).

Dexamethasone treatment is currently practiced for various pathologies afflicting the inner ear. The positive effect of Dexamethasone is attributed to it's anti ROS activity and it's capability to up-regulate cochlear anti ROS enzymes.

In order to reach higher inner ear concentration of the drug while avoiding it's undesirable systemic side-effects, Intratympanic (IT) delivery of Dexamethasone became vastly used in the last decades for the treatment of sudden sensorineural hearing loss and Meniere's disease.

Dexamethasone inserted IT, diffuse across the round window into the inner ear perilymph where it exerts its therapeutic effects.

The investigators review of the literature yielded three animal studies which examined the protective effect of IT dexamethasone in the prevention of cisplatin-induced hearing loss. These studies demonstrated promising results pointing to the potential for IT dexamethasone in the prevention of cisplatin ototoxicity in humans.

The purpose of this study is to examine possible protective effect of IT dexamethasone on cisplatin-induced hearing loss, in humans.

The study hypothesis is that IT dexamethasone treatment would prevent cisplatin-induced hearing loss.

DETAILED DESCRIPTION:
Prevention of Cisplatin-Induced Hearing Loss by Intratympanic Dexamethasone Treatment.

Introduction:

Cisplatin is a widely used chemotherapeutic agent for the treatment of various malignant neoplasms, including testicular, ovarian, bladder, cervix uteri, head and neck and lung cancers 1-4.

Dose limiting side effects of Cisplatin include nephrotoxicity, neurotoxicity and ototoxicity. While nephrotoxicity can be diminished or controlled with hydration therapy there are no known cure or preventive treatments available for neurotoxicity and ototoxicity 2,4.

Cisplatin-associated ototoxicity is characterized by bilateral, symmetric progressive and usually irreversible sensorineural hearing loss. The hearing impairment is dose related, cumulative and takes place within hours to days from the administration of cisplatin 1-4. The reported incidence of cisplatin-induced hearing loss is variable. Schweitzer calculated from a large number of studies an average incidence of 62% with a range from 11 to 97% 5-6. Damage from cisplatin initially affects the outermost row of outer hair cells located at the cochlear basal turn, which codes hearing at the high frequency range. Further insult affects the remaining rows of outer hair cells, inner hair cells, and supporting cells. The pattern of destruction proceeds from the basal turn towards the more apical regions of the cochlea, with increasing impact on hearing acuity in lower frequencies 7.

Cisplatin induces cochlear toxicity by the production of reactive oxygen species (ROS) on one hand and depletion of antioxidant enzymes on the other hand. This leads to lipid, protein and nucleic acids peroxidation with destruction of various cell organs and apoptosis 4,7,8.

Various chemoprotectants have been suggested to ameliorate cisplatin-induced ototoxcity. These include sodium thiosulfate, amifostine, diethyldithiocarbamate, 4-methylthiobenzoic acid, D- and L-methionine, N-acetylcysteine, and glutathione ester. The mechanisms of action include direct antioxidant activity and maintenance of glutathione levels 2,4. Unfortunately, systemic delivery of many of these agents have been found to inhibit the tumoricidal effects of cisplatin and/or have toxicities or unknown effects in humans 2,9.

Abundant corticosteroids receptors were demonstrated within the mouse critical inner ear structures suggesting active role of these compounds in inner ear homeostasis 10. Dexamethasone has been reported to up-regulate cochlear anti ROS enzymes activity in various small mammals animal models2,3,11.

Dexamethasone treatment is currently practiced for various pathologies afflicting the inner ear in which ROS are involved in immediate or delayed ischemia-reperfusion mechanism of injury. These include sudden sensorineural hearing loss, noise-induced hearing loss, salicylate and aminoglycoside ototoxicity 2.

The above discussion suggests rationale for the prevention of cisplatin ototoxicity by Dexamethasone.

Intratympanic (IT) delivery of drugs is a contemporary method based on the diffusion of the active remedy across the round window into the inner ear where it exerts its therapeutic effects 12-14. This method allows for high inner ear concentration when compared to oral or parenteral administration while avoiding the undesirable systemic side-effects 12.

IT administration of steroids is vastly used in the last decades for the treatment of sudden sensorineural hearing loss and Meniere's disease. 2,3,12 Currently employed techniques for IT drug delivery include trans-tympanic membrane injection into the middle ear cavity either directly or through a tympanostomy; placing a wick attached to the round window niche which is suggested to facilitate better administration of the drug to the target organ; implantation of a round window microcatheter connected to a micro-pump for continuous drug delivery. Experimental IT strategies include the application of various hydrogels and nanoparticles as drug carriers, and direct delivery of medication to the inner ear via osmotic pumps and reciprocating perfusion systems 12.

Our review of the literature yielded three animal studies which examined the protective effect of IT dexamethasone in the prevention of cisplatin-induced hearing loss. These studies demonstrated promising results pointing to the potential for IT dexamethasone in the prevention of cisplatin ototoxicity in humans. Daldal et al carried a controlled study in the guinea pig model. The study groups were treated by IT dexamethasone either before or after intra-peritoneal injections of cisplatin, one control group had cisplatin injections alone and the second control group was given only IT dexamethasone. IT dexamethasone caused no cochlear damage as evaluated by distortion product otoacoustic emissions (DPOAEs). Cisplatin caused significant decrease in DPOAEs amplitudes and SNR values, while both IT dexamethasone treated groups demonstrated significant protection from cisplatin ototoxicity 11. Hill et al evaluated ABR click and tone burst evoked thresholds in mice receiving intra-peritoneal cisplatin. In each animal one ear was treated by IT dexamethasone while the second ear had IT saline injection and served as a control. The results showed significant protection for the click, 8 and 16 kHz threshold shifts in the IT dexamethasone treated ears 3. Paksoy et al employed similar ABR evaluations to examine the potential otoprotective effect of IT dexamethasone in cisplatin treated rats. While significant thresholds elevations were demonstrated in the cisplatin treated rats, IT dexamethasone preserved ABR responses 2.

We could not find any previously published study that examined the role of IT dexamethasone in the prevention of cisplatin-induced ototoxicity in humans.

The purpose of this study is to examine possible protective effect of IT dexamethasone on cisplatin-induced hearing loss, in humans.

Our study hypothesis is that IT dexamethasone treatment would prevent cisplatin-induced hearing loss.

Patients and Methods:

The study design is a prospective cohort controlled research. The participants would be 30 consecutive patients suffering from a neoplastic disease for which the treatment protocol includes cisplatinum not previously delivered to them. The cumulative cisplatin dose would be at least 300mg divided to treatment sessions and dosages as dictated by the oncologist.

After receiving an explanation about the study goals and methods, candidates for participation in the study would sign an informed consent.

Baseline evaluation would include detailed history with emphasis on previous or existing ear disease, microscopic otoscopy, pure tone, speech and impedance audiometry, and Distortion Product Otoacoustic Emissions (DPOAEs) testing. This test specifically evaluates the functioning of the cochlear outer hair cells which are the primary target organ for cisplatin ototoxicity. It has been previously shown that decreased signal-to-noise ratio (SNR) of the otoacoustic emissions precedes the appearance of the audiological pure tone threshold shift and identify sub-clinical hearing loss.15 Exclusion criteria would include the followings: age < 18 years; existing or previous pathology of the external or middle ear avoiding IT drug delivery or the performance of DPOAEs testing; retrocochlear hearing loss; Meniere's disease; Autoimmune Inner Ear Disease; fluctuating hearing loss; history of sudden sensory neural hearing loss; previous radiation therapy to the head and neck region; baseline average pure tone audiometry thresholds for 500-3000 Hz and 4000-8000 Hz greater than 40 dB; average SNR below 6 dB for DPOAEs f2 frequencies 500-3000 Hz and 4000-8000 Hz.

Under topical anesthesia of Emla cream (mixture of lidocaine 2.5% and prilocaine 2.5%), 0.7ml of Dexamethasone Phosphate 10mg/ml would be injected unilaterally to the middle ear using 25 gauge spinal needle. The injected side would serve as the study ear while the contralateral side would be the control ear. The ear receiving the treatment would be randomly chosen using a computerized "randomizer"16. The trans-tympanic membrane injection would take place at the posterior inferior quadrant of the ear drum facing the round window niche. The patient would be instructed to lie down for 20 minutes after the injection with the treated side up and to avoid swallowing or coughing. These measures are taken to allow maximal contact of the Dexamethasone solution with the round window membrane while minimizing medication loss via the Eustachian tube. Intratympanic Dexamethasone would be delivered immediately prior to each cisplatin treatment as maximal level of the medication in the scala tympani is anticipated 1 hour post injection 10,17,18 while the maximal perilymph concentration of cisplatinum after intravenous injection in the guinea pig model is reached after 20 minutes19.

Pure tone, speech and impedance audiometry and DPOAEs would be recorded prior to the first cisplatinum administration and before each consecutive treatment. The final testing would take place 7 days after the last treatment session in which the cumulative dose of 300mg was achieved.

The following parameters would be compared between the study and control ears for the baseline and consecutive examinations: Pure tone average thresholds for 500-3000 and 4000-8000 Hz; DPOAEs SNR averages for 500-3000 and 4000-8000 f2 frequencies.

Normal distribution of the results would be examined by the Shapiro-Wilk test. The comparisons between the study and control ears for the baseline and consecutive evaluations would be done using the Student's paired two-tailed t-test. Longitudinal changes in pure tone audiometry thresholds and DPOAEs SNR would be evaluated by repeated measures ANOVA.

Sample size calculation was based on the following parameters: The event rate for cisplatinum-induced sensorineural hearing loss is 60% 6; each patient serves as his own control when one ear is treated and the hearing level is compared to that of the untreated ear; A successful treatment is defined as preventing at least third of the anticipated hearing loss in the study population; the desired statistical power is 80% with p<0.05.

Taking the above parameters into consideration the calculated required sample size is 30 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from a neoplastic disease for which the treatment protocol includes cisplatinum not previously delivered to them.
* The cumulative cisplatin dose would be at least 300mg.

Exclusion Criteria:

* Age < 18 years.
* Existing or previous pathology of the external or middle ear avoiding IT drug delivery or the performance of DPOAEs testing.
* Retrocochlear hearing loss.
* Meniere's disease.
* Autoimmune Inner Ear Disease.
* fluctuating hearing loss.
* History of sudden sensory neural hearing loss.
* Previous radiation therapy to the head and neck region.
* Baseline average pure tone audiometry thresholds for 500-3000 Hz and 4000-8000 Hz greater than 40 dB.
* Average SNR below 6 dB for DPOAEs f2 frequencies 500-3000 Hz and 4000-8000 Hz.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Examine possible protective effect of IT dexamethasone on cisplatin-induced hearing loss. Hearing assessment would include:pure tone, speech and impedance audiometry, and Distortion Product Otoacoustic Emissions (DPOAEs) testing. | Two years
  Distortion Product Otoacoustic Emissions (DPOAEs) testing is a test that specifically evaluates the functioning of the cochlear outer hair cells which are the primary target organ for cisplatin ototoxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Tal M Marshak, MD, Principal Investigator — Clalit Health Services
Locations (1):
- Clalit Health Services, Haifa, Israel